CLINICAL TRIAL: NCT05549297
Title: Phase 2/3 Randomized Study of Tebentafusp as Monotherapy and in Combination With Pembrolizumab Versus Investigator's Choice in HLA-A*02:01-positive Participants With Previously Treated Advanced Melanoma (TEBE-AM)
Brief Title: Tebentafusp Regimen Versus Investigator's Choice in Previously Treated Advanced Melanoma (TEBE-AM)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMCgp100-203
Record Dates: First submitted 2022-08-26; First posted 2022-09-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Advanced Melanoma
Keywords: Melanoma; IMCgp100; Tebentafusp; Cutaneous Melanoma; Immunotherapy; gp100; TCR; Pembrolizumab; Bispecific T cell receptor fusion protein; ImmTAC (Immune-mobilizing monoclonal T-cell receptor Against Cancer); Immune mobilizing monoclonal T cell receptor against cancer; KIMMTRAK; Acral Melanoma; Mucosal Melanoma; Blue Nevus; anti-PDL1; checkpoint therapy
MeSH Terms: conditions — Melanoma; Nevus, Blue | interventions — tebentafusp; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Tebentafusp Monotherapy (Experimental): Participants receive tebentafusp as single agent.
  Interventions: Drug: Tebentafusp
- Arm B: Tebentafusp + Pembrolizumab (Experimental): Participants receive tebentafusp in combination with pembrolizumab.
  Interventions: Drug: Tebentafusp with Pembrolizumab
- Arm C: Investigator's Choice (Experimental): Participants receive investigator's choice of therapy.
  Interventions: Drug: Investigators Choice

INTERVENTIONS:
Drug: Tebentafusp — Soluble gp100-specific T cell receptor with anti-CD3 scFV
  Arms: Arm A: Tebentafusp Monotherapy
Drug: Tebentafusp with Pembrolizumab — Soluble gp100-specific T cell receptor with anti-CD3 scFV in combination with pembrolizumab
  Arms: Arm B: Tebentafusp + Pembrolizumab
Drug: Investigators Choice — Investigators choice of therapy
  Arms: Arm C: Investigator's Choice

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tebentafusp-based regimens, including tebentafusp monotherapy and in combination with anti-PD1 vs investigator choice (including clinical trials of investigational agents, salvage therapy per local standard of care [SoC], best supportive care [BSC] on protocol survivor follow up) in patients with advanced non-ocular melanoma.

DETAILED DESCRIPTION:
This is a phase 3 (as upon conversion to phase 3 there were no changes to the arms listed herein), multicenter, open-label study to evaluate the efficacy and safety of tebentafusp as monotherapy (Arm A) and in combination with pembrolizumab (Arm B) compared with standard of care or best supportive care (Arm C) in participants with non-ocular advanced melanoma who have progressed on a prior anti-PD(L)1 regimen, received an approved anti-CTLA4 regimen and, if the participant has a BRAF mutation, a prior BRAF tyrosine kinase inhibitor (TKI) regimen.

ELIGIBILITY:
Inclusion Criteria:

* HLA-A*02:01-positive
* unresectable Stage III or Stage IV non-ocular melanoma
* archival tumor tissue sample or a newly obtained biopsy of a tumor lesion not previously irradiated has been provided.
* measurable or non-measurable disease per RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* If applicable, must agree to use highly effective contraception
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the Informed Consent (ICF) and protocol
* Must agree to provide protocol specified samples for biomarker analyses.

Exclusion Criteria:

* Pregnant or lactating women
* diagnosis of ocular or metastatic uveal melanoma
* history of a malignant disease other than those being treated in this study
* ineligible to be retreated with pembrolizumab due to a treatment-related AE
* known untreated or symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis
* previous severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb)
* active autoimmune disease requiring immunosuppressive treatment
* clinically significant cardiac or pulmonary disease or impaired cardiac function
* known psychiatric or substance abuse disorders
* received prior treatment with a licensed or investigative Immune-mobilizing monoclonal T-cell receptor Against Cancer (ImmTAC) medication or who have not completed adequate washout from prior medications.
* received chemotherapy or biological cancer therapy (excluding anti-PD(L)1 mAb, ipilimumab, and BRAF TKI regimen) within 14 days of first dose
* received cellular therapies within 90 days of study intervention
* ongoing Common Terminology Criteria for Adverse Events(CTCAE) Grade ≥ 2 clinically significant who in the opinion of the investigator could affect the outcome of the study
* received systemic treatment with steroids or any other immunosuppressive drug within 2 weeks of first dose
* have not progressed on treatment with an anti-PD(L)1 mAb
* have not received prior treatment with an approved anti-CTLA-4 mAb
* a BRAF V600 mutation, who have not received a prior BRAF/MEK TKI regimen
* currently participating or have participated in a study of an investigational agent or using an investigational device within 30 days of the first dose
* known history of chronic viral infections such as hepatitis B virus (HBV) or hepatitis C virus (HCV)
* known clinically significant pulmonary or cardiac disease or impaired lung or cardiac function
* Out of range Laboratory values
* history of allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to ~4 years
  OS is the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Change from Baseline in Circulating Tumor DNS (ctDNA) | Up to ~9 weeks
  Change from baseline in ctDNA will be assessed.
Number of participants with ≥1 adverse event (AE) | Up to ~4 years
  Number of participants with AEs.
Number of participants with ≥1 serious adverse event (SAEs) | Up to ~4 years
  Number of participants with SAEs.
Number of participants with dose interruptions, reductions, and discontinuations from study therapy due to AEs | Up to ~4 years
  Number of participants with tolerability issues.
Number of participants with Grade ≥2 cytokine release syndrome (CRS) | Up to ~4 years
  CRS based on American Society for Transplantation and Cellular Therapy (ASTCT) criteria.
Responses to the EORTC Core Quality of Life (EORTC-QLQ-C30) | At designated time points up to ~4 years
  Participant-reported quality of life.
Responses to the European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) | At designated time points up to ~4 years
  Participant-reported quality of life.
Plasma Concentration of Tebentafusp | At designated time points up to ~4 years
  Plasma concentration of tebentafusp.
Number of participants with anti-tebentafusp antibodies | At designated time points up to ~4 years
  The number of participants with anti drug antibodies (ADA) to tebentafusp.

CONTACTS AND LOCATIONS:
Locations (71):
- United States (17):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Northwell Health Cancer Institute - Zuckerberg Cancer Center, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Medical Oncology Clinic, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Houston Methodist Hospital/Houston Methodist Cancer Center, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (4):
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - Gallipoli Medical Research Foundation (GMRF), Greenslopes, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Alfred Health, Melbourne, Victoria
- Austria (4):
  - LKH - Universitaetsklinikum Graz, Graz
  - Kepler Universitätsklinikum, Linz
  - Universitatsklinik fur Innere Medizin 3, Salzburg
  - AKH - Medizinische Universität Wien, Vienna
- Belgium (3):
  - Cliniques Universitaires Sain-Luc, Brussels
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
- Princess Margaret Hospital, Toronto, Ontario, Canada
- France (6):
  - Centre Leon Berard, Lyon, Cedex
  - Institute Claudius Regaud, Toulouse, Cedex
  - Institut Gustave Roussy, Villejuif, Cedex
  - CHU de Bordeaux - Hopital Saint Andre, Bordeaux
  - Hopital de la Timone [Recruiting], Marseille
  - Hopital Saint Lous - APHP, Paris
- Germany (11):
  - Universitaetsklinikum Schleswig-Holstein, Schleswig, Kiel
  - Charité - Campus Charité Mitte, Berlin
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Johannes Wesling Klinikum Minden, Minden
  - LMU-Campus Innenstadt, München
  - Universitaetsklinikum Tübingen, Tübingen
- Italy (5):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Instituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Azienda Ospedaliera di Perugia Ospedale S. Maria della Misericordia, Perugia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - A.O.U Senese Policlinico Santa Maria alle Scotte, Siena
- Poland (4):
  - Centrum Onkologii im. prof. F. Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne (UCK) - Klinika Onkologii i Radioterapii, Gdansk
  - Szpital Kliniczny im.Heliodora Swiecickiego Uniwersytetu Medycznego im.K. Marcinkowskiego w Poznaniu, Poznan
  - Narodowy Instytut Onkologii-im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinico de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital General Universitario de Valencia, Valencia
- Switzerland (2):
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitaetsspital Zurich, Zurich
- United Kingdom (8):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - Leeds General Infirmary, Leeds
  - Guys & St Thomas' NHS Foundation Trust, London
  - Sarah Cannon Research Institute UK, London
  - Royal Marsden Hospital - Chelsea, London
  - Mount Vernon Cancer Center, Middlesex
  - Royal Marsden Hospital - Sutton, Sutton